CLINICAL TRIAL: NCT00875160
Title: An Open-Label Study to Assess the Pharmacokinetics, Safety, and Pharmacodynamics of Repeated Doses of Orally Administered AT2101 in Adult Patients With Type 1 Gaucher Disease
Brief Title: A Study in Type 1 Gaucher Patients to Evaluate the Pharmacokinetics, Safety and Pharmacodynamics of AT2101
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Subject Recruitment
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Eugene Schneider, MD, Medical Director, Clinical Research, Amicus Therapeutics
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAU-CL-104
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2010-08-19 (Estimated); Status verified 2010-08

CONDITIONS: Type 1 Gaucher Disease
MeSH Terms: conditions — Gaucher Disease | interventions — AT2101

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AT2101 (Experimental)
  Interventions: Drug: AT2101

INTERVENTIONS:
Drug: AT2101 — 225mg (nine 25mg capsules total dose) to be taken by mouth every day for 9 days (Study Days 1, 3-10)

SUMMARY:
This is an open-label study designed to assess if AT2101 is safe in patients with Gaucher disease and how AT2101 gets through the body after it is taken by mouth. The study is being offered to adult patients with type 1 Gaucher disease who are currently receiving a stable dose of enzyme replacement therapy (ERT) with imiglucerase. During the study, subjects will not be receiving ERT (up to 35 days).

The study consists of a screening period (~14 days), a treatment period (12 days) and a follow-up period (7 days after last dose). At two points in the study, subjects will be housed in an in-patient treatment facility for 3 days/2 nights to accommodate all necessary blood draws.

DETAILED DESCRIPTION:
While on the study, subjects will be required to refrain from consuming the following foods and beverages:

* Caffeine: 24 hours before admission and throughout the in-patient stay;
* Alcohol: 48 hours before admission and throughout the in-patient stay. A maximum of 2 units/day will be allowed during the out-patient part of the study (1 unit of alcohol = wind (125mL)=spirits(25mL)=beer (284mL);
* Vitamins: throughout the in-patient periods.

Subjects will also be restricted to taking medications or herbal products during the study except if the Principal Investigator permits.

Subjects will not engage in strenuous activity at any time during the in-patient periods.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of type 1 Gaucher disease with a documented gene mutation;
* Clinically stable and on a stable dose of ERT for at least 2 years before study entry, with no changes to dose level or regimen in the last 6 months;
* Willing to stop ERT for the duration of the study;
* Male or female between the ages of 18 to 65 inclusive;
* All subjects of reproductive potential are required to practice an acceptable method of contraception;
* All subjects must have a body mass index of less than 30; and
* Provide written informed consent to participate in the study.

Exclusion Criteria:

* A clinically significant disease, severe complications from Gaucher disease, or serious intercurrent illness that may preclude participation in the study in the opinion of the Investigator;
* During the screening/wash out period, any clinically significant findings, based on physical exam, medical history review, lab assessment, vital sign assessment and/or other significant finding which would compromise the safety of the subject, or preclude the subject from completing the study as deemed by the Investigator;
* Partial or total splenectomy;
* History of pulmonary hypertension or Gaucher-related lung disease;
* History of allergy or sensitivity to the study drug or any excipients, including any prior serious allergic reaction to iminosugars;
* Screening or Day 1 (before dosing) 12-lead ECG demonstration QTc >450 msec in males or >470 in females;
* Pregnant or breast-feeding;
* Current/recent drug or alcohol abuse within the past 12 months;
* Treatment with any investigational product, including investigational forms of ERT, in the 90 days before study entry;
* Treatment in the previous 90 days with any drug known to have a well-defined potential for toxicity to a major organ;
* Presence or sequelae of gastrointestinal, liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs; or
* Subject is otherwise unsuitable for the study in the opinion of the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To evaluate single-dose and multiple-dose pharmacokinetics of isofagomine following the oral administration of AT2101 in patients with type 1 Gaucher disease | Multiple times for up to three days following Day 1 and Day 10

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of oral AT2101 administered in patients with type 1 Gaucher disease | Daily
To evaluate the pharmacodynamic effect of WBC GCase of oral AT2101 administered in patients with type 1 Gaucher disease. | Days 1, 5 & 7 (optional), 10 and 17

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Schneider, MD, Study Director — Amicus Therapeutics
Locations (2):
- Comprehensive Phase One, Miramar, Florida, United States
- Guy's Drug Research Unit, London, United Kingdom